CLINICAL TRIAL: NCT01798563
Title: Functional Connectivity of the Motor Network in Two Major Subtypes of Parkinson Disease
Brief Title: Functional Connectivity Parkinson Disease
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 10-1311
Record Dates: First submitted 2012-12-11; First posted 2013-02-26 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Tremor Dominant PD: Volunteers with predominantly tremor-related motor symptoms of PD
- Postural Instability & Gait Difficulty PD: Volunteers with primarily walking & balance-related motor symptoms of PD.
- Healthy Controls: Healthy volunteers consisting of people of same age as PD volunteers, w/o a diagnosis of PD.

SUMMARY:
In this study the investigators are looking at two subtypes of Parkinson Disease (PD); "tremor-dominant" (TD) and postural imbalance and gait disorder (PIGD). This study will use magnet resonance imaging (MRI) to see how the brain reacts while resting and doing a finger-tapping task while on and off PD medication. This study will look at the differences between the two sub-types of PD and healthy volunteers.

The investigators will test the hypothesis that connectivity at rest within the motor cortex and between the motor cortex and motor-associated regions such as the supplementary motor area and the pre motor cortex will not be as strong in PIGD compared to TD (increased activity and functional connectivity in TD group)

ELIGIBILITY:
Inclusion Criteria:

* English as their primary language
* Patients with Parkinson disease and healthy controls will be enrolled
* Parkinson patients must be on a dopaminergic medication (levodopa or dopamine agonist) and on a stable dose over the prior month

Exclusion Criteria:

* If unable to provide informed consent
* Pregnancy
* Excess of 300lbs
* Claustrophobia
* Metal in body
* Untreated neurological or psychiatric condition, who are delusional or have hallucinations, with cognitive impairment (MOCA<26), with a history of head injury sufficient to cause a concussion, or with significant systemic medical diseases (e.g. heart failure, liver failure, kidney failure, poorly controlled diabetes, etc.)
* Healthy control subjects will be excluded if taking any type of dopaminergic or anti-dopaminergic medication
* Subjects who are unable to demonstrate understanding of the study procedures and risks will be excluded

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with PD according to UK Brain Bank Criteria will be recruited from the UCD Neurology clinic. Controls will be recruited from spouses and from the community
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2011-06; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Correlation coefficients between nodes of the motor network at rest and during a tapping motor task. | At time of MRI scan: 12 or more hours after their last dose of dopaminergic medication.
  A measure of the correlation coefficients between nodes of the motor network at rest and during a tapping motor task between the "OFF" and "ON" dopaminergic medication states in the two motor subtype PD patients.
Correlation coefficients between nodes of the motor network at rest and during a tapping motor task. | At time of 2nd MRI scan: 1 to 3 hours after taking their usual dose(s) dopaminergic medication(s).
  A measure of the correlation coefficients between nodes of the motor network at rest and during a tapping motor task between the "OFF" and "ON" dopaminergic medication states in the two motor subtype PD patients.
Second level contrast between Parkinson Disease (PD) and Healthy Controls (HC). | At time of MRI scan: 12 or more hours after their last dose of dopaminergic medication.
  Differences in connectivity as measured by correlation coefficients between nodes of the motor network at rest and during a tapping motor task in PD patients of two motor subtypes and matched healthy controls.

SECONDARY OUTCOMES:
Task-related whole-brain activations. | At time of MRI scan, 12 or more hours after their last dose of dopaminergic medication.
  Secondary outcome measures include task-related whole-brain activations as assessed by changes in blood oxygen-dependent (BOLD) contrast during functional magnetic resonance imaging (fMRI) scanning.
Task-related whole-brain activations. | At time of 2nd MRI scan, 1 to 3 hours after taking their usual dose(s) dopaminergic medication(s).
  Secondary outcome measures include task-related whole-brain activations as assessed by changes in blood oxygen-dependent (BOLD) contrast during functional magnetic resonance imaging (fMRI) scanning.
Connectivity between other motor and non-motor brain regions during the tasks. | At time of MRI scan,12 or more hours after their last dose of dopaminergic medication.
  Secondary outcome measures include measuring the connectivity between other motor and non-motor brain regions during the tasks.
Correlations of brain activity and functional connectivity to structural connectivity measures and behavioral and clinical assessments | At time of MRI scan. 12 or more hours after their last dose of dopaminergic medication.
  Secondary outcome measures include a measure of the correlations of brain activity and functional connectivity to structural connectivity measures as well as behavioral and clinical assessments.
Correlations of brain activity and functional connectivity to structural connectivity measures and behavioral and clinical assessments | At time of 2nd MRI scan. 1 to 3 hours after taking their usual dose(s) dopaminergic medication(s).
  Secondary outcome measures include a measure of the correlations of brain activity and functional connectivity to structural connectivity measures as well as behavioral and clinical assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Berman, MD, MS, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No